CLINICAL TRIAL: NCT02443545
Title: Long-term Safety and Efficacy Study of Ferriprox® for the Treatment of Transfusional Iron Overload in Patients With Sickle Cell Disease or Other Anemias
Brief Title: Long-term Safety and Efficacy of Ferriprox® in Iron Overloaded Patients With Sickle Cell Disease or Other Anemias
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recommendation by DSMB, which felt that sufficient data had been obtained
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Organization: Chiesi Canada Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA38-EXT
Record Dates: First submitted 2015-05-05; First posted 2015-05-14 (Estimated); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Iron Overload; Sickle Cell Disease; Other Anemias
Keywords: Iron overload; Sickle cell disease; Deferiprone; Ferriprox; Iron chelation
MeSH Terms: conditions — Iron Overload; Anemia, Sickle Cell | interventions — Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Deferiprone 3 years (Experimental): Patients in this group are those who were randomized to the deferiprone arm in study LA38-0411, and hence will receive deferiprone for a total of 3 years (1 year in the initial study plus 2 years in the extension study).
  Interventions: Drug: Deferiprone
- Group 2: Deferiprone 2 years (Experimental): Patients in this group are those who were randomized to the deferoxamine arm in study LA38-0411, and hence will receive deferiprone for 2 years (both of them in the extension study).
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone
  Other Names: Ferriprox tablets; Ferriprox oral solution

SUMMARY:
This is a long-term follow-up to an earlier study, LA38-0411. Its purpose is to gather more information about the safety and efficacy of deferiprone in patients with sickle cell disease or other anemias who suffer from iron overload caused by regular blood transfusions.

DETAILED DESCRIPTION:
Deferiprone (brand name Ferriprox®) is an iron chelator that is approved in the United States and over 60 other countries for the treatment of iron overload in patients with thalassemia, when other treatments are inadequate. This study has been designed to evaluate the long-term efficacy, safety, and tolerability of deferiprone to treat iron overload in patients who have sickle cell disease or other anemias.

Only patients who have completed an earlier study, LA38-0411, are eligible to enroll in this one.

ELIGIBILITY:
Inclusion Criteria:

1. Completed study LA38-0411
2. Females of childbearing potential must have a negative pregnancy test result at Visit 1. In addition, if applicable, they must:

   * Use an effective method of contraception according to local requirements, during the study and within 30 days following their last dose of study medication, OR
   * Have had a tubal ligation (supporting evidence required), OR
   * Have had a hysterectomy (supporting evidence required), OR
   * Participate in a non-heterosexual lifestyle, OR
   * Have a male sexual partner who has been sterilized (supporting evidence required)
3. Fertile heterosexual males and/or their partners must agree to use an effective method of contraception during the study and for 30 days following the last dose of study medication
4. All patients and/or their authorized legal representatives must provide signed and dated written informed consent prior to the first study intervention, and assent will be obtained from patients who are considered to be minors. Patients must be able to adhere to study restrictions, appointments, and evaluation schedules.

Exclusion Criteria:

1. Plan to participate in another clinical trial at any time from the day of enrollment until 30 days post-treatment in the current study
2. For only those patients who were treated with deferoxamine in study LA38-0411 (Group 2): Presence of any medical condition (including clinically significant laboratory abnormalities, such as ALT (alanine aminotransferase) ≥ 5 x ULN or creatinine ≥ 2 x ULN), psychological condition, or psychiatric condition which in the opinion of the investigator would cause participation in the study to be unwise.
3. Pregnant, breastfeeding, or planning to become pregnant during the study period.
4. Treatment failure after 1 year on deferiprone which in the investigator's judgment indicates the need for the patient to be started on a different iron chelator

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kwiatkowski, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (13):
- United States (5):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - The Children's Hospital of Philadephia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Hospital for Sick Kids, Toronto, Ontario, Canada
- Egypt (4):
  - Zagazig University, Alexandria
  - Ain Shams University, Cairo
  - Cairo University, Cairo
  - Pediatric Hospital of Cairo University, Cairo
- Asser Central Hospital, Abhā, Saudi Arabia
- United Kingdom (2):
  - Barts and The London, London
  - Evelina Children's Hospital, London

REFERENCES:
- [Derived] Elalfy MS, Hamdy M, El-Beshlawy A, Ebeid FSE, Badr M, Kanter J, Inusa B, Adly AAM, Williams S, Kilinc Y, Lee D, Fradette C, Rozova A, Temin NT, Tricta F, Kwiatkowski JL. Deferiprone for transfusional iron overload in sickle cell disease and other anemias: open-label study of up to 3 years. Blood Adv. 2023 Feb 28;7(4):611-619. doi: 10.1182/bloodadvances.2021006778. PMID 36018224

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Deferiprone 3 Years: Patients in this group are those who were randomized to the deferiprone arm in study LA38-0411 (NCT02041299), and hence will receive deferiprone for a total of 3 years (1 year in the initial study plus 2 years in the extension study)..
  Deferiprone
- Group 2: Deferiprone 2 Years: Patients in this group are those who were randomized to the deferoxamine arm in study LA38-0411 (NCT02041299), and hence will receive deferiprone for 2 years (both of them in the extension study).
  Deferiprone
Period: Overall Study
Arm/Group | Group 1: Deferiprone 3 Years | Group 2: Deferiprone 2 Years
Started | 89 | 45
Completed | 50 | 26
Not Completed | 39 | 19
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Protocol Violation | 8 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Termination of study | 20 | 11

BASELINE CHARACTERISTICS:
Groups:
- Deferiprone: All patients in this study received deferiprone
Arm/Group | Deferiprone
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 133
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 114
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 5
  Canada | 2
  United States | 14
  Egypt | 109
  United Kingdom | 4
Liver iron concentration at baseline [Mean (Standard Deviation); unit: mg iron per gram of liver dry weight] — Liver iron concentration is measured by MRI. A value > 7 milligrams of iron per gram of liver dry weight (mg/g dw) is indicative of iron overload.
  mg iron per gram of liver dry weight | 14.93 (7.61)
Cardiac iron at baseline [Mean (Standard Deviation); unit: milliseconds] — Cardiac iron is measured by MRI. A value < 20 ms is indicative of iron overload.
  milliseconds | 32.69 (17.66)
Serum ferritin level at baseline [Mean (Standard Deviation); unit: micrograms per liter] — Normal levels of serum ferritin are under 300 µg/L for females and under 400 µg/L for males.
  micrograms per liter | 3894 (2591)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events
Description: Number of patients with at least one adverse event (AE) of any type; number of patients with at least one serious adverse event, and number of patients who withdrew from the study due to an AE
Time Frame: From the first day of the study until the last study visit (Week 104 or early termination)
Population: Safety population (all enrolled patients who took at least one dose of study drug)
Measure: Count of Participants; unit: Participants
Arm/Group | Deferiprone
Number analyzed (Participants) | 134
Participants
  Number of patients with any type of adverse event | 104
  Number of patients with a serious adverse event | 35
  Number of patients who discontinued due to an AE | 2

2. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC)
Description: LIC was measured by MRI, in units of mg of iron per gram of liver (dry weight). The change from baseline in LIC was determined for three different periods of exposure to deferiprone: one year, two years, and three years.
Time Frame: One year, two years, and three years after the start of deferiprone therapy
Population: Intent-to-Treat (ITT) population (patients who received at least one dose of study drug and had a baseline and at least one post-baseline efficacy assessment). LIC data for one year of exposure to deferiprone were obtained from 129 patients, data for two years from 112 patients, and data for three years from 59 patients.
Measure: Mean (Standard Deviation); unit: mg of iron per gram of liver dry weight
Arm/Group | Deferiprone
Number analyzed (Participants) | 129
mg of iron per gram of liver dry weight
  Change from baseline in LIC after 1 year | -2.64 (4.64)
  Change from baseline in LIC after 2 years: number analyzed (Participants) | 112
  Change from baseline in LIC after 2 years | -3.91 (6.38)
  Change from baseline in LIC after 3 years: number analyzed (Participants) | 59
  Change from baseline in LIC after 3 years | -6.64 (7.72)
Statistical Analysis 1: Comparison: Deferiprone; Change from baseline after 1 year of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in LIC was significantly different from 0; p = 0.0000, t-test, 2 sided
Statistical Analysis 2: Comparison: Deferiprone; Change from baseline after 2 years of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in LIC was significantly different from 0; p = 0.0000, t-test, 2 sided
Statistical Analysis 3: Comparison: Deferiprone; Change from baseline after 3 years of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in LIC was significantly different from 0; p = 0.0000, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Cardiac MRI T2*
Description: The change from baseline in cardiac MRI T2* was determined for three different periods of exposure to deferiprone: one year, two years, and three years
Time Frame: One year, two years, and three years after the start of deferiprone therapy
Population: ITT population. Cardiac MRI T2* data for one year of exposure to deferiprone were obtained from 121 patients, data for two years from 110 patients, and data for three years from 58 patients.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Deferiprone
Number analyzed (Participants) | 121
milliseconds
  Change from baseline in cardiac iron after 1 year | 1.02 (19.65)
  Change from baseline in cardiac iron after 2 years: number analyzed (Participants) | 110
  Change from baseline in cardiac iron after 2 years | 1.00 (21.18)
  Change from baseline in cardiac iron after 3 years: number analyzed (Participants) | 58
  Change from baseline in cardiac iron after 3 years | 0.98 (24.53)
Statistical Analysis 1: Comparison: Deferiprone; Change from baseline after 1 year of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in MRI T2* was significantly different from 0; p = 0.3146, t-test, 2 sided
Statistical Analysis 2: Comparison: Deferiprone; Change from baseline after 2 years of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in MRI T2* was significantly different from 0; p = 0.9454, t-test, 2 sided
Statistical Analysis 3: Comparison: Deferiprone; Change from baseline after 3 years of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in MRI 2* was significantly different from 0; p = 0.4336, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: The change from baseline in serum ferritin (SF) was determined for three different periods of exposure to deferiprone: one year, two years, and three years.
Time Frame: One year, two years, and three years after the start of deferiprone therapy
Population: ITT population. Serum ferritin data for one year of exposure to deferiprone were obtained from 125 patients, data for two years from 96 patients, and data for three years from 55 patients.
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Deferiprone
Number analyzed (Participants) | 125
micrograms per liter
  Change from baseline in SF after 1 year | -1 (1986)
  Change from baseline in SF after 2 years: number analyzed (Participants) | 96
  Change from baseline in SF after 2 years | -771 (2171)
  Change from baseline in SF after 3 years: number analyzed (Participants) | 55
  Change from baseline in SF after 3 years | -1016 (3617)
Statistical Analysis 1: Comparison: Deferiprone; Change from baseline after 1 year of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in serum ferritin was significantly different from 0; p = 0.9952, t-test, 2 sided
Statistical Analysis 2: Comparison: Deferiprone; Change from baseline after 2 years of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in serum ferritin was significantly different from 0; p = 0.0008, t-test, 2 sided
Statistical Analysis 3: Comparison: Deferiprone; Change from baseline after 3 years of deferiprone therapy; Test type: Other — One-sample t-test, to determine whether the change from baseline in serum ferritin was significantly different from 0; p = 0.0420, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to end of study (up to 2 years)
Arm/Group | Deferiprone
All-Cause Mortality (participants affected / at risk) | 1/134
Serious Adverse Events (participants affected / at risk) | 35/134
Other Adverse Events (participants affected / at risk) | 99/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=134)
Agranulocytosis (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 12 (15)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 19 (42)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (6)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2)
Propionibacterium infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 3 (3)
Medical device repositioning (Surgical and medical procedures) | 1 (1)
Splenectomy (Surgical and medical procedures) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferiprone (N=134)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 17 (39)
Abdominal pain (Gastrointestinal disorders) | 26 (44)
Vomiting (Gastrointestinal disorders) | 9 (12)
Pyrexia (General disorders) | 33 (50)
Nasopharyngitis (Infections and infestations) | 17 (28)
Pharyngitis (Infections and infestations) | 10 (15)
Upper respiratory tract infection (Infections and infestations) | 9 (12)
Neutrophil count decreased (Investigations) | 16 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (51)
Bone pain (Musculoskeletal and connective tissue disorders) | 35 (97)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (33)
Headache (Nervous system disorders) | 12 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (28)

LIMITATIONS AND CAVEATS:
The trial was terminated early upon recommendation of the Data and Safety Monitoring Board (DSMB), which felt that sufficient information had been obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02443545/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT02443545/SAP_001.pdf